CLINICAL TRIAL: NCT05856682
Title: Pre-incision Versus Lapaorscopic-assisted Transversus Abdominis Plane (TAP) and Rectus Sheath Block for Post-Cholecystectomy Pain Management: A Randomized Controlled Trial
Brief Title: Pre-incision Versus Lapaorscopic-assisted Transversus Abdominis Plane (TAP) and Rectus Sheath Block for Post-Cholecystectomy Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Patel Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Kanwal Nisa, Kanwal Nisa, Patel Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PatelHospital
Record Dates: First submitted 2023-04-21; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: randomized, prospective, double blinded
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded study : participants and person assessing the post operative pain will be blinded to both the control and intervention group, person performing TAP block will not be assessing the outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-incision TAP (PITAP) and Rectus Sheath block (Active Comparator): Pre-incision TAP block and Rectus sheath block will be performed after induction of anesthesia, just after prep and drape by Blind double pop technique by Anesthetist/Anesthesia trainee.Site of rectus block will be Bilaterally 3 cm lateral to Umblicus and 3cm lateral to midpoint between xiphisternum and umbilicus . Site of TAP block will be Immediate right subcostal region , 3 cm medially to mid axillary line The intervention and the control group will receive TAP block and rectus sheath block with Rupivacaine (3mg/kg). 1 ampule is of 10 ml and consists of 50mg /10ml, maximum dose will be 300mg. will use a of minimum volume of solution 50ml which will be made by 3 ampules of Rupivacaine and it will be diluted to a total of 20ml of injectate( distilled water )which is then divided between the four rectus block sites (5ml each) and one TAP block site(30ml ).
  Interventions: Procedure: Laparoscopic-assisted TAP block(LATAP) and Rectus Sheath block
- Laparoscopic-assisted TAP block(LATAP) and Rectus Sheath block (Active Comparator): Laparoscopic -assisted TAP and rectus sheath block will be performed after insertion of optical port By Surgeon /surgery trainee.Site of rectus block will be Bilaterally 3 cm lateral to Umblicus and 3cm lateral to midpoint between xiphisternum and umbilicus . Site of TAP block will be Immediate right subcostal region , 3 cm medially to mid axillary line The intervention and the control group will receive TAP block and rectus sheath block with Rupivacaine (3mg/kg). 1 ampule is of 10 ml and consists of 50mg /10ml, maximum dose will be 300mg. will use a of minimum volume of solution 50ml which will be made by 3 ampules of Rupivacaine and it will be diluted to a total of 20ml of injectate( distilled water )which is then divided between the four rectus block sites (5ml each) and one TAP block site(30ml each).
  Interventions: Procedure: Laparoscopic-assisted TAP block(LATAP) and Rectus Sheath block

INTERVENTIONS:
Procedure: Laparoscopic-assisted TAP block(LATAP) and Rectus Sheath block — Laparoscopic -assisted TAP and rectus sheath block will be performed after insertion of optical port By Surgeon /surgery trainee. • Site of rectus block will be Bilaterally 3 cm lateral to Umblicus and 3cm lateral to midpoint between xiphisternum and umbilicus . Site of TAP block will be anterior to the midaxillary line between the costal margin and iliac crest bilaterally.
  Other Names: Pre-incision TAP (PITAP) and Rectus Sheath block

SUMMARY:
The goal of this clinical trial is to compare pre-incision vs laparoscopic assisted Transversus abdominis plane and rectus sheath block in patients undergoing laparoscopic cholecystectomy. The main question it aims to answer is:

• if the effectiveness of TAP and rectus sheath block varies according to whether it is performed pre-incisional (pre emptive) or intraoperatively under Laparoscopic vision for laparoscopic cholecystectomies.

Participants will be assessed for pain at 3,6,12, and 24 hrs after surgery. Researchers will compare pain score between Laparoscopic-assisted TAP block(LATAP) and Rectus Sheath block vs Pre-incision TAP (PITAP ) .

DETAILED DESCRIPTION:
INTRODUCTION:

Every year Over 13 million Laparoscopic procedures are performed globally. In the USA, 90% of the cholecystectomies are performed with the laparoscopic technique

* Laparoscopic cholecystectomy is the gold standard in many health centers as it is less invasive compared to open cholecystectomy.
* Good post-operative pain control, not only prevents post-operative complications but is also essential for early ambulation and return to daily routine. It is important to keep side effects minimum besides pain relieve. Therefore pre-emptive wound analgesia has been popularized. Preemptive analgesia(for eg: TAP block) is defined as an anti-nociceptive treatment that is initiated before the surgical procedure in order to reduce the sensitization (occurs because of transmission of pain signals evoked by tissue damage) of the peripheral and central pain pathways. Some analyses have shown no beneficial effect(4) whereas some have failed to reach a final conclusion regarding efficacy of pre-emptive analgesia.
* For post-laparoscopic pain management ,a multimodal approach with non-steroidal anti-inflammatory drugs, opioids and loco-regional techniques have been recommended . The Transversus Abdominis Plane (TAP) block is an analgesia technique that is loco-regional ,consists of infiltrating a local anesthetic solution between the plane of the Transversus abdominis muscle and the internal oblique muscle.
* TAP block has gradually become an alternative postoperative analgesia technology and it was described in 2001 by Rafi. . Several techniques are currently used to deliver TAP blocks, including blinded double pop technique, ultrasound-guided and laparoscopic-assisted approaches. The latter was first described in 2011 by Chetwood et al. while performing laparoscopic nephrectomies . The advantages of this technique include ease of performance, less dependency on specialized skill set or equipment, time efficient, less risk of visceral injury and avoidance of intraperitoneal local anaesthetic infiltration .

RATIONALE: Many studies have demonstrated the therapeutic benefit of laparoscopic-assisted TAP block in initial post-operative pain management in comparision with periportal local anaesthetic infiltration for patients undergoing elective laparoscopic procedures(for eg; for laparoscopic hernia repair). To the best of our knowledge, there is a paucity of data since laparoscopic-assisted TAP block has not been utilized or evaluated prospectively to see if the effectiveness of TAP block varies according to whether it is performed pre-incisional (pre emptive) or intraoperatively under Laparoscopic vision for laparoscopic cholecystectomies. Moreover, the rectus sheath block in conjunction with TAP block has not been evaluated before.

OBJECTIVE :

To compare the mean post-operative pain score at (3, 6, 12, 24 hours) with pre-incision versus laparoscopic-assisted Transversus Abdominis Plane (TAP) and Rectus sheath block in patients undergoing Laparoscopic cholecystectomy at a tertiary care hospital.

HYPOTHESIS : Post-Cholecystectomy pain control after Laparoscopic-assisted TAP block is not inferior to pain control after pre-incisional TAP block.

OPERATIONAL DEFINITIONS :

Transversus abdominis plane(TAP block): It is a regional analgesia technique which involves the injection of a local anesthetic solution into a plane between the internal oblique muscle and transversus abdominis muscle. Since the thoracolumbar nerves originating from the T6 to L1 spinal roots run into this plane and supply sensory nerves to the antero-lateral abdominal wall , the local anesthetic spread in this plane can block the neural afferents and provide analgesia to the antero-lateral abdominal wall.

Rectus sheath block : It is a method of trunk analgesia most useful for midline surgical procedures at or above the umbilicus. Local anesthetic is injected at the lateral edge of the rectus sheath where branches of the intercostal nerves enter. Instillation of local anesthetic bilaterally between the rectus muscle and the posterior sheath provides midline analgesia for several dermatomes around the injection site.

Pain score (visual analogue scale):

The Visual Analogue Scale (VAS) is the standard tool for rating of pain - either patient's own rating or rated by the health care worker. The visual analog scale is a straight line from 1 to 10 with one end meaning no pain and the other end meaning the worst pain. A patient marks a point on the line that matches the intensity of pain he or she feels.

MATERIALS AND METHODS:

* STUDY DESIGN: Double blinded, Randomized controlled trial
* SETTINGS: The study will be conducted at the department of General Surgery, Patel hospital Karachi.
* DURATION OF STUDY: After ERC approval, minimum Six months or till the sample size is achieved.
* RANDOMIZATION: Computer generated randomization table with blocks of four. Co-ordinator of HEC will have the table.
* BLINDING: Double blinded (Patient, Person assessing post-operative pain will be blinded to the both groups).
* INTERVENTION GROUP: Laparoscopic-assisted TAP block(LATAP) and Rectus Sheath block
* CONTROL GROUP: Pre-incision TAP (PITAP) block by Anesthesist.
* SAMPLE SIZE : In each arm, 112 patients.
* SAMPLE CALCULATION METHOD: Calculated using WHO software.
* Power set as =90%
* Confidence interval =95%
* Level of significance = 5%
* SAMPLING TECHNIQUE: Purposive, non probability

DATA COLLECTION PROCEDURE:

* Study will be started after approval by the institutional ethical committee.
* Detailed history, examination and relevant investigations of patients will be performed.
* Informed and written consent will be taken.
* Proforma will be filled for patients undergoing planned surgery fulfilling the inclusion criteria .
* Anesthesia will be standardized in all patients.
* All patients will receive paracetamol 1000 mg and nalbuphine 0.15mg/kg after induction of anaesthesia.
* Both the procedures will be performed by either Resident(having experience of procedure) or consultant himself/herself.
* Syringes will be prepared by one of the research team member for each patient in a designated sterile area on the day of surgery..
* Pre-incision TAP block and Rectus sheath block will be performed after induction of anesthesia, just after prep and drape by Blind double pop technique by Anesthetist/Anesthesia trainee
* Laparoscopic -assisted TAP and rectus sheath block will be performed after insertion of optical port By Surgeon /surgery trainee
* Site of rectus block will be Bilaterally 3 cm lateral to Umblicus and 3cm lateral to midpoint between xiphisternum and umbilicus . Site of TAP block will be Immediate right subcostal region , 3 cm medially to mid axillary line .
* The intervention and the control group will receive TAP block and rectus sheath block with Rupivacaine (3mg/kg). 1 ampule is of 10 ml and consists of 50mg /10ml, maximum dose will be 300mg. We will use a of minimum volume of solution 50ml which will be made by 3 ampules of Rupivacaine and it will be diluted to a total of 20ml of injectate( distilled water )which is then divided between the four rectus block sites (5ml each) and one TAP block site(30ml).
* Needle used for the blocks will be of 25guage and tip of the needle will be blunted by gentle tapping on metallic surface. Syringe will be of 50ml .
* Timings of PITAP AND LATAP will be noted in seconds by putting the timer on at the start of the procedures when anesthesia/surgery team calls the procedure on and by putting the timer off ,when they calls the procedure off.
* Peritoneal entry will be seen under laparoscopic vision. For LATAP ,entry would be labelled when tip of needle will be seen piercing peritoneum and for PITAP any erythema or bleed at the site of entry seen under laparoscopic vision.
* Visceral entry will be seen under laparoscopic vision for both LATAP and PITAP.
* Diet will be Regular and started after 6 hours of the surgery.
* Ambulation will be started as soon as patient is awake .
* Antibiotics (cefazolin 1gm ,q8hrly) will be prescribed post-operatively to contaminated surgery.
* Patient-controlled analgesia(PCA) will be given in the post-operative period for all patients for rescue analgesia and explained to them pre-operatively. On having pain, as per need , Patient will press the button on a pump that is connected to IV catheter. Patient will receive a preset dose of Nalbuphine 2mg.
* Pain assessment will be measured using the visual analogue scale (0-10). Pain will be assessed at both rest and coughing (reflect pain induced by physical activity) at 3,6,12, and 24 hrs after surgery by an observer blinded to both intervention and control group.

DATA ANALYSIS plan:

SPSS (ver. 16) will be used for data analysis. Confounding and effect modifying variables i.e. age, sex, diabetes are analyzed by multiple linear regression. For Data that will follow normality Independent sample T test will be applied, for data that will not follow normality Mann- whitney u test will be applied. P-value of less than 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 to 75 years, both genders, Elective Laparoscopic Cholecystectomies, American Society of Anesthesiologists (ASA) physical status I & II, Give consent.

Exclusion Criteria:

* o History of allergy , hypersentivity or contraindication to Rupivacaine, nalbuphine ,Paracetamol.

  * Local skin allergy
  * Laparoscopic converted to open
  * Previous open upper abdominal or midline surgeries
  * Diagnosis Of "Chronic Pain Syndrome"
  * Known Alcohol Or Substance Abuse Within The Last 6 Months
  * Anti-psychotic, antidepressants, steroids use
  * Multiple procedures planned under single GA
  * Pregnancy
  * Unable to understand i.e. deaf, language barrier, mentally incapacitated
  * Coagulopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain changes | 3,6,12,24 hrs post-operatively
  post operative chnage of pain score assessment at 3,6,12,24 hrs at resting and coughing. Pain score will be assessed using VAS score

SECONDARY OUTCOMES:
Rescue analgesia need | Post operatively at 3,6,12,24hrs
  if any additional anlagesia is required , nalbuphine 2mg IV as per need will be used via PCA pump.
Visceral Injury | at the time of surgery
  if any viscera is damage during TAP and rectus sheath block in both groups
Peritoneal injury | at the time of surgery
  • Peritoneal entry will be seen under laparoscopic vision. For LATAP ,entry would be labelled when tip of needle will be seen piercing peritoneum and for PITAP any erythema or bleed at the site of entry seen under laparoscopic vision.
TAP and rectus sheath block timings | at the time of surgery
  comparsion of timings between both groups ,• Timings of PITAP AND LATAP will be noted in seconds by putting the timer on at the start of the procedures when anesthesia/surgery team calls the procedure on and by putting the timer off ,when they calls the procedure off.

CONTACTS AND LOCATIONS:
Locations (1):
- Patel Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amreek F, Hussain SZM, Mnagi MH, Rizwan A. Retrospective Analysis of Complications Associated with Laparoscopic Cholecystectomy for Symptomatic Gallstones. Cureus. 2019 Jul 16;11(7):e5152. doi: 10.7759/cureus.5152. PMID 31523579
- [Background] Csikesz NG, Singla A, Murphy MM, Tseng JF, Shah SA. Surgeon volume metrics in laparoscopic cholecystectomy. Dig Dis Sci. 2010 Aug;55(8):2398-405. doi: 10.1007/s10620-009-1035-6. Epub 2009 Nov 13. PMID 19911275
- [Background] Ortiz J, Rajagopalan S. A review of local anesthetic techniques for analgesia after laparoscopic surgery. J Minim Invasive Surg Sci. 2014;3:e11310
- [Background] Tsai HC, Yoshida T, Chuang TY, Yang SF, Chang CC, Yao HY, Tai YT, Lin JA, Chen KY. Transversus Abdominis Plane Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:8284363. doi: 10.1155/2017/8284363. Epub 2017 Oct 31. PMID 29226150
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] Elamin G, Waters PS, Hamid H, O'Keeffe HM, Waldron RM, Duggan M, Khan W, Barry MK, Khan IZ. Efficacy of a Laparoscopically Delivered Transversus Abdominis Plane Block Technique during Elective Laparoscopic Cholecystectomy: A Prospective, Double-Blind Randomized Trial. J Am Coll Surg. 2015 Aug;221(2):335-44. doi: 10.1016/j.jamcollsurg.2015.03.030. Epub 2015 Mar 27. PMID 25899736
- [Background] Chetwood A, Agrawal S, Hrouda D, Doyle P. Laparoscopic assisted transversus abdominis plane block: a novel insertion technique during laparoscopic nephrectomy. Anaesthesia. 2011 Apr;66(4):317-8. doi: 10.1111/j.1365-2044.2011.06664.x. No abstract available. PMID 21401554
- [Background] Mughal A, Khan A, Rehman J, Naseem H, Waldron R, Duggan M, Khan W, Barry K, Khan IZ. Laparoscopic-assisted transversus abdominis plane block as an effective analgesic in total extraperitoneal inguinal hernia repair: a double-blind, randomized controlled trial. Hernia. 2018 Oct;22(5):821-826. doi: 10.1007/s10029-018-1819-8. Epub 2018 Sep 1. PMID 30173291
- [Background] Chapter 57 - Rectus Sheath Block, Editor(s): Andrew T. Gray, Atlas of Ultrasound-Guided Regional Anesthesia (Third Edition),Elsevier, 2019,Pages 249-258,ISBN 9780323509510.
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- See also: Related Info — http://idataresearch.com/over-13-million-laparoscopic-procedures-are-performed-globally-every-year/